CLINICAL TRIAL: NCT04978129
Title: Examining Motivations for and Quality of Alcohol and Marijuana Protective Behavior Strategy Use: Improving Prevention of Hazardous Young Adult Substance Use
Brief Title: Enhancing Quality in Protective Strategies
Acronym: EQUIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melissa Lewis, PhD, Professor of School of Social Work, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7R34AA028730-04 (NIH); 7R34AA028730-04 (NIH)
Record Dates: First submitted 2021-06-24; First posted 2021-07-27 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Health Risk Behaviors; Risk Reduction Behavior
MeSH Terms: conditions — Health Risk Behaviors; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online and Text Message Intervention (Experimental): Participants randomized to the intervention will receive a link to the online intervention following baseline completion. The online and Text Message intervention, and its delivery, will be designed and adapted based on the results of the formative focus groups and cognitive interviews and is meant to be non-confrontational in tone, seeks to increase motivation to increase the quality use of PBS and decrease motivations for non-use of PBS. Intervention participants will receive personalized PBS Text Messages 3x per week (based on self-selections from the interactive online intervention) for 8 consecutive weeks timed to occur on a random weekday as well as Friday and Saturday.
  Interventions: Behavioral: Online and Text Messaging Intervention
- Assessment Only Control (No Intervention): The assessment only control condition will not receive any intervention content during the 8-week period of data collection, but will complete baseline, 2-month, and daily surveys according to the same schedule as the intervention group in order to assess event-level PBS use, PBS non-use, alcohol and marijuana use, CAM and SAM use, and related consequences for up to 24 days over an 8-week period.

INTERVENTIONS:
Behavioral: Online and Text Messaging Intervention — The online and TM intervention, and its delivery, will be designed and adapted based on the results of the formative focus groups and cognitive interviews and is meant to be non-confrontational in tone, seeks to increase motivation to increase the quality use of PBS and decrease motivations for non-use of PBS.
  Arms: Online and Text Message Intervention

SUMMARY:
The most successful young adult alcohol or marijuana interventions involve the provision of accurate, nonjudgmental personalized feedback, but notably the inclusion and effectiveness of protective behavioral strategies (PBS) content is inconsistent. Moreover, active components of brief interventions are not well understood, and findings have been inconclusive regarding whether PBS mediates intervention efficacy of college student personalized feedback interventions (PFIs), with only some studies showing evidence of mediation. One possible reason for these findings is that investigators often do not know young adults' motivations for using (or not using) PBS or the quality of PBS use across individuals or across drinking occasions. The proposed study will provide an in-depth examination of which PBS young adults are motivated to use (including implementation quality) and reasons that young adults may or may not use PBS. Understanding why young adults are choosing not to use PBS on specific occasions or do not engage in effective or high-quality PBS use on certain occasions has significant clinical implications, whereby interventions may need to spend more time increasing motivations to use PBS in an effective manner or work on reducing perceived barriers (i.e., reasons individuals are not using PBS). Clinicians may then be better able to work with young adults in various settings to reduce or prevent excessive alcohol and marijuana use and related consequences. The proposed research has high potential for making a substantial impact on the field and public health (particularly as more states permit legal access to marijuana for those over 21) as it will address a problem of high importance (alcohol and marijuana use) by being the first to develop and refine a PBS intervention that specifically focuses on motivations for alcohol and marijuana PBS use and non-use as well as quality of use, which is an overlooked aspect of current PBS-related intervention approaches. The development of more efficacious interventions to reduce the proportion of young adults who engage in excessive alcohol use and who experience consequences is a key priority of the NIAAA. Related, development of more effective interventions to reduce risk from marijuana use is an area of great importance for the NIDA.

DETAILED DESCRIPTION:
The majority of young adults who use both alcohol and marijuana do so simultaneously. Simultaneous Alcohol and Marijuana (SAM) use is defined as using alcohol and marijuana at the same time so that their effects overlap. Individuals who engage in Concurrent Alcohol and Marijuana (CAM) use are often characterized as those who report both alcohol and marijuana use within the same time period (e.g., past month, past week). An increasing body of literature has documented CAM and SAM use on a given day among young adults. Event-level findings show SAM use is associated with increased risk for consequences, compared to marijuana use alone or CAM use. Given that the investigators' focus in this application is on daily-level substance use behaviors, the investigators define CAM use as using both substances on the same day, but not so that their effects overlap. Interventions should focus on reducing drinking as well as drinking that occurs in conjunction with marijuana use to provide a more comprehensive evaluation of intervention efficacy. The proposed research in this application will develop and test a novel online and text message (TM) protective behavioral strategies (PBS) intervention to reduce alcohol, marijuana, CAM, and SAM use and related negative consequences among young adults.

One way interventions could prevent or reduce alcohol- and marijuana-related consequences is by promoting the use of PBS, which are behaviors that individuals can use to limit consequences and/or reduce substance use. PBS are often incorporated into brief interventions or TM interventions in the form of skills training. Despite the empirical support for including PBS content in brief interventions, findings have been inconclusive regarding whether PBS mediate intervention efficacy among college students. One possible explanation is that skills-based PBS interventions prematurely focus on "how" to use PBS, but not "why" PBS might be used or used with high quality. Research is needed to determine motivations for when and why young adults may or may not decide to use PBS to reduce harm while using alcohol and/or marijuana, which can then enable investigators to better address these motivations in brief interventions. Research has yet to examine how alcohol and marijuana PBS use on a given day relates to an individual's use of alcohol alone or marijuana alone in comparison to CAM or SAM use. The proposed study will fill these critical gaps by identifying the extent to which motivations for PBS use and nonuse (marijuana or alcohol) and quality of PBS use (degree of effectiveness or degree of implementation) differ when using alcohol alone versus concurrently or simultaneously with marijuana. The overall goal of this research is to inform a pilot study of a newly developed alcohol and marijuana PBS intervention. The proposed research will (1) collect pilot data to establish feasibility and acceptability and test the interactive online and TM PBS intervention (baseline, 2-month) while also (2) collecting event-level data to examine daily-level associations among PBS motivation/quality, PBS use and non-use, alcohol and/or marijuana use, and negative consequences with a focus on how PBS may differ on CAM or SAM use days compared to alcohol-only days.

Aim 1: Examine motivations for alcohol and marijuana PBS use (and non-use of PBS) as well as quality of PBS use among young adults (ages 18-24) who use both alcohol and marijuana. The present study will conduct online focus groups (10 groups, N=10 individuals per group) and cognitive interviews (N=10) to determine why young adults use or do not use specific PBS related to alcohol and/or marijuana use. Focus groups will address how PBS use or motivations to avoid consequences may differ by gender (male, female, non-binary). Focus groups and cognitive interviews will discuss the level of quality in which PBS are used and various contexts in which PBS may or may not be used. Discussions will consider use of either substance alone on a given day as well as SAM or CAM use on a given day and will include ways in which the motivations and quality of PBS could be incorporated into an online and TM PBS intervention, as well as elicit feedback on mock intervention material. Using an exploratory sequential mixed methods design, an iterative process of focus groups and cognitive interviews will inform the development and delivery of the intervention to be tested in the pilot study (Aim 2). Aim 1 is not a clinical trial.

Aim 2: Conduct a pilot study with young adults (N=200; ages 18-24), who typically use alcohol and marijuana at least two days per week, to determine feasibility, acceptability, and preliminary effect sizes (to inform a future R01 application). Participants will be randomized to either the intervention or wait-list control. The intervention is a brief interactive online intervention focusing on self-selected alcohol and marijuana PBS messages and motives for using alcohol- and marijuana-related PBS and includes intervention content delivered via TMs three days a week (random day, Friday, Saturday) over eight consecutive weekends. All participants will report PBS use, motivations for PBS use (and non-use), quality of PBS use, readiness to change, and alcohol and marijuana use in morning surveys timed to occur the day after the intervention TMs for those in the intervention group. The proposed research in this application will provide an in-depth understanding of young adults' PBS use and has potential to develop a more efficacious intervention for these co-occurring or simultaneous alcohol and marijuana behaviors. Aim 2 is the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-24
2. Live in Texas
3. Valid email address
4. Own a cell phone with text messaging capabilities
5. Okay with receiving messages
6. Typically drink at least 2 days a week
7. Typically use marijuana at least 2 days a week
8. Report having at least 1 alcohol-related and 1 marijuana-related consequence in the past month
9. Report being in contemplation or action stage based on readiness to change scale for alcohol or marijuana (i.e., not in precontemplation stage)
10. If female, not pregnant or trying to become pregnant
11. Not currently in treatment for alcohol or substance use
12. Willing to participate in either online focus group or online cognitive interview (Phase I) or pilot study with daily morning surveys (Phase II), and willing to receive study notifications on phone (e.g., survey reminders) [Phase II]
13. Their device must meet the system requirements to participate in the online focus group or cognitive interview (have iOS 8.0 or later, Android 4.0x, or later, or have another video-enabled device) [Phase I]

Exclusion Criteria:

1. Not meeting inclusion criteria
2. Unwillingness to participate
3. Failure to provide consent
4. Providing inconsistent responses (e.g., age), and
5. Having already participated in the study as identified by overlap or consistency in email addresses, contact information, and demographics.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Lewis, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
A select number of researchers will have access to unidentified participant data at the close of the study.

REFERENCES:
- [Background] National Institute on Alcohol Abuse and Alcoholism (2019). Planning alcohol interventions using NIAAA's College Alcohol Intervention Matrix (CollegeAIM). Bethesda, MD: National Institutes of Health, (NIH Publication No. 19-AA-8017, Updated December 2019).
- [Background] Miller, W. R., & Rollnick, S. (2013). Motivational interviewing: Helping people change (3rd ed.). New York, NY: Guilford Press.
- [Background] Gaume J, McCambridge J, Bertholet N, Daeppen JB. Mechanisms of action of brief alcohol interventions remain largely unknown - a narrative review. Front Psychiatry. 2014 Aug 26;5:108. doi: 10.3389/fpsyt.2014.00108. eCollection 2014. PMID 25206342
- [Background] Reid AE, Carey KB. Interventions to reduce college student drinking: State of the evidence for mechanisms of behavior change. Clin Psychol Rev. 2015 Aug;40:213-24. doi: 10.1016/j.cpr.2015.06.006. Epub 2015 Jun 24. PMID 26164065
- [Background] Subbaraman MS, Kerr WC. Simultaneous versus concurrent use of alcohol and cannabis in the National Alcohol Survey. Alcohol Clin Exp Res. 2015 May;39(5):872-9. doi: 10.1111/acer.12698. PMID 25872596
- [Background] Egan KL, Cox MJ, Suerken CK, Reboussin BA, Song EY, Wagoner KG, Wolfson M. More drugs, more problems? Simultaneous use of alcohol and marijuana at parties among youth and young adults. Drug Alcohol Depend. 2019 Sep 1;202:69-75. doi: 10.1016/j.drugalcdep.2019.07.003. Epub 2019 Jul 6. PMID 31319362
- [Background] Lipperman-Kreda S, Gruenewald PJ, Grube JW, Bersamin M. Adolescents, alcohol, and marijuana: Context characteristics and problems associated with simultaneous use. Drug Alcohol Depend. 2017 Oct 1;179:55-60. doi: 10.1016/j.drugalcdep.2017.06.023. Epub 2017 Jul 20. PMID 28755540
- [Background] Martens MP, Taylor KK, Damann KM, Page JC, Mowry ES, Cimini MD. Protective behavioral strategies when drinking alcohol and their relationship to negative alcohol-related consequences in college students. Psychol Addict Behav. 2004 Dec;18(4):390-3. doi: 10.1037/0893-164X.18.4.390. PMID 15631613
- [Background] Pedersen ER, Hummer JF, Rinker DV, Traylor ZK, Neighbors C. Measuring Protective Behavioral Strategies for Marijuana Use Among Young Adults. J Stud Alcohol Drugs. 2016 May;77(3):441-50. doi: 10.15288/jsad.2016.77.441. PMID 27172576
- [Background] Murphy JG, Dennhardt AA, Skidmore JR, Borsari B, Barnett NP, Colby SM, Martens MP. A randomized controlled trial of a behavioral economic supplement to brief motivational interventions for college drinking. J Consult Clin Psychol. 2012 Oct;80(5):876-86. doi: 10.1037/a0028763. Epub 2012 Jun 4. PMID 22663899
- [Background] Riggs NR, Conner BT, Parnes JE, Prince MA, Shillington AM, George MW. Marijuana eCHECKUPTO GO: Effects of a personalized feedback plus protective behavioral strategies intervention for heavy marijuana-using college students. Drug Alcohol Depend. 2018 Sep 1;190:13-19. doi: 10.1016/j.drugalcdep.2018.05.020. Epub 2018 Jun 23. PMID 29960918
- [Background] Cadigan JM, Martens MP, Dworkin ER, Sher KJ. The Efficacy of an Event-Specific, Text Message, Personalized Drinking Feedback Intervention. Prev Sci. 2019 Aug;20(6):873-883. doi: 10.1007/s11121-018-0939-9. PMID 30054777
- [Background] Lewis MA, Cadigan JM, Cronce JM, Kilmer JR, Suffoletto B, Walter T, Lee CM. Developing Text Messages to Reduce Community College Student Alcohol Use. Am J Health Behav. 2018 Jul 1;42(4):70-79. doi: 10.5993/AJHB.42.4.7. PMID 29973312
- [Background] Miller MB, Leffingwell T, Claborn K, Meier E, Walters S, Neighbors C. Personalized feedback interventions for college alcohol misuse: an update of Walters & Neighbors (2005). Psychol Addict Behav. 2013 Dec;27(4):909-20. doi: 10.1037/a0031174. Epub 2012 Dec 31. PMID 23276309
- [Background] Collins RL, Parks GA, Marlatt GA. Social determinants of alcohol consumption: the effects of social interaction and model status on the self-administration of alcohol. J Consult Clin Psychol. 1985 Apr;53(2):189-200. doi: 10.1037//0022-006x.53.2.189. No abstract available. PMID 3998247
- [Background] Johnston, L. D., O'Malley, P. M., Bachman, J. G., & Schulenberg, J. E. (2012). Monitoring the Future national results on adolescent drug use: Overview of key findings, 2011. Ann Arbor: Institute for Social Research, The University of Michigan.
- [Background] Babor, T. F., Higgins-Biddle, J. C., Saunders, J. B., Monteiro, M. G. (2001). AUDIT- The alcohol use disorders identification test: guidelines for use in primary care (Research Report No. (WHO/MSD/MSB/01.6a). http://whqlibdoc.who.int/hq/2001/WHO_MSD_MSB_01.6a.pdf
- [Background] Read JP, Kahler CW, Strong DR, Colder CR. Development and preliminary validation of the young adult alcohol consequences questionnaire. J Stud Alcohol. 2006 Jan;67(1):169-77. doi: 10.15288/jsa.2006.67.169. PMID 16536141
- [Background] Treloar H, Martens MP, McCarthy DM. The Protective Behavioral Strategies Scale-20: improved content validity of the Serious Harm Reduction subscale. Psychol Assess. 2015 Mar;27(1):340-6. doi: 10.1037/pas0000071. Epub 2015 Jan 5. PMID 25558969
- [Background] Litt, D. M. & Lewis, M. A. (2016). An Examination of Protective Behavioral Strategies, Motivations for Strategy Selection, and Alcohol Use Among Young Adults. Poster presented at the Association for Behavioral and Cognitive Therapies, New York.
- [Background] Bravo AJ, Pearson MR, Stevens LE, Henson JM. Weighing the Pros and Cons of Using Alcohol Protective Behavioral Strategies: A Qualitative Examination among College Students. Subst Use Misuse. 2018 Nov 10;53(13):2190-2198. doi: 10.1080/10826084.2018.1464026. Epub 2018 Apr 30. PMID 29708460
- [Background] Heather, N., & Hönekopp, J. (2008). A revised edition of the Readiness to Change Questionnaire [Treatment Version]. Addiction Research & Theory, 16(5), 421-433. https://doi.org/10.1080/16066350801900321
- [Background] Lee CM, Kilmer JR, Neighbors C, Atkins DC, Zheng C, Walker DD, Larimer ME. Indicated prevention for college student marijuana use: a randomized controlled trial. J Consult Clin Psychol. 2013 Aug;81(4):702-9. doi: 10.1037/a0033285. Epub 2013 Jun 10. PMID 23750464
- [Background] Simons JS, Dvorak RD, Merrill JE, Read JP. Dimensions and severity of marijuana consequences: development and validation of the Marijuana Consequences Questionnaire (MACQ). Addict Behav. 2012 May;37(5):613-21. doi: 10.1016/j.addbeh.2012.01.008. Epub 2012 Jan 14. PMID 22305645
- [Background] Stephens RS, Roffman RA, Fearer SA, Williams C, Picciano JF, Burke RS. The Marijuana Check-up: reaching users who are ambivalent about change. Addiction. 2004 Oct;99(10):1323-32. doi: 10.1111/j.1360-0443.2004.00832.x. PMID 15369571
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Pedersen ER, Huang W, Dvorak RD, Prince MA, Hummer JF; (The Marijuana Outcomes Study Team). The Protective Behavioral Strategies for Marijuana Scale: Further examination using item response theory. Psychol Addict Behav. 2017 Aug;31(5):548-559. doi: 10.1037/adb0000271. Epub 2017 Jul 13. PMID 28703616
- [Background] Brown SA, Myers MG, Lippke L, Tapert SF, Stewart DG, Vik PW. Psychometric evaluation of the Customary Drinking and Drug Use Record (CDDR): a measure of adolescent alcohol and drug involvement. J Stud Alcohol. 1998 Jul;59(4):427-38. doi: 10.15288/jsa.1998.59.427. PMID 9647425
- [Background] Schafer J, Brown SA. Marijuana and cocaine effect expectancies and drug use patterns. J Consult Clin Psychol. 1991 Aug;59(4):558-65. doi: 10.1037//0022-006x.59.4.558. PMID 1918560
- [Background] Substance Abuse and Mental Health Services Administration. Enhancing Motivation for Change in Substance Use Disorder Treatment. Treatment Improvement Protocol (TIP) Series No. 35. SAMHSA Publication No. PEP19-02-01-003. Rockville, MD: Substance Abuse and Mental Health Services Administration, 2019
- [Background] Johnston, L. D., O'Malley, P. M., Miech, R. A., Bachman, J. G., & Schulenberg, J. E. (2015). Monitoring the Future national survey results on drug use: 1975-2014: Overview, key findings on adolescent drug use: 1975-2014 [PDF File]. Ann Arbor: Institute for Social Research, The University of Michigan. https://deepblue.lib.umich.edu/handle/2027.42/137913.
- [Background] Brooke, J. (1996). SUS: A quick and dirty usability scale. In Jordan PW, Thomas B, Weerdmeester BA, McClelland IL (Eds.), Usability evaluation in industry (pp. 189-194). London, England: Taylor & Francis.
- [Background] Brooke, J. (2013). SUS: A retrospective. Journal of Usability Studies, 8(2), 29-40.
- [Background] Sauro, J. (2011). A practical guide to the system usability scale: Background, benchmarks, & best practices. Denver, CO: Measuring Usability LLC.
- [Background] Danielson CK, McCauley JL, Gros KS, Jones AM, Barr SC, Borkman AL, Bryant BG, Ruggiero KJ. SiHLEWeb.com: Development and usability testing of an evidence-based HIV prevention website for female African-American adolescents. Health Informatics J. 2016 Jun;22(2):194-208. doi: 10.1177/1460458214544048. Epub 2014 Aug 28. PMID 25167865
- [Background] Li, X., Lewis, M. A., Fairlie, A. M., & Mun, E. Y. (2019, June). Participants come back to see web-delivered personalized feedback aimed at reducing alcohol-related risky sexual behavior among young adults. Poster presented at the annual meeting of the Research Society on Alcoholism, Minneapolis, MN.
- [Background] Shrier LA, Burke PJ, Kells M, Scherer EA, Sarda V, Jonestrask C, Xuan Z, Harris SK. Pilot randomized trial of MOMENT, a motivational counseling-plus-ecological momentary intervention to reduce marijuana use in youth. Mhealth. 2018 Jul 30;4:29. doi: 10.21037/mhealth.2018.07.04. eCollection 2018. PMID 30148142
- [Background] Lewis MA, Litt DM, King KM, Fairlie AM, Waldron KA, Garcia TA, LoParco C, Lee CM. Examining the ecological validity of the prototype willingness model for adolescent and young adult alcohol use. Psychol Addict Behav. 2020 Mar;34(2):293-302. doi: 10.1037/adb0000533. Epub 2019 Nov 21. PMID 31750697
- [Background] Stephens RS, Roffman RA, Curtin L. Comparison of extended versus brief treatments for marijuana use. J Consult Clin Psychol. 2000 Oct;68(5):898-908. PMID 11068976
- [Background] White, H. R., Labouvie, E. W., Papadaratsakis, V. (2005). Changes in substance use during the transition to adulthood: A comparison of college students and their noncollege age peers. Journal of Drug Issues, 35(2), 281-306. doi:10.1177/002204260503500204
- [Background] Linden-Carmichael AN, Van Doren N, Masters LD, Lanza ST. Simultaneous alcohol and marijuana use in daily life: Implications for level of use, subjective intoxication, and positive and negative consequences. Psychol Addict Behav. 2020 May;34(3):447-453. doi: 10.1037/adb0000556. Epub 2020 Jan 23. PMID 31971426
- [Derived] Lewis MA, Litt DM, Fairlie AM, Kilmer JR, Kannard E, Resendiz R, Walker T. Investigating Why and How Young Adults Use Protective Behavioral Strategies for Alcohol and Marijuana Use: Protocol for Developing a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 19;11(4):e37106. doi: 10.2196/37106. PMID 35438642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Texas state using a variety of recruitment methods. Individuals were invited to complete an online eligibility survey for participation in a randomized clinical trial to test the effect of an online and text message personalized feedback intervention. Recruitment/enrollment and data collection period went from August 2023 to October 2024.
Period: Overall Study
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Started | 83 | 79
Completed | 78 | 75
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online and Text Message Intervention | Assessment Only Control | Total
Number analyzed (Participants) | 83 | 79 | 162
Age, Continuous [Mean (Full Range); unit: Years] | 22.18 [18 to 24] | 22 [18 to 24] | 22.09 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 104
  Male | 30 | 28 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race. The number of participants represents those who provided data for this outcome measure.
  Participants
    American Indian or Alaska Native | 4 | 5 | 9
    Asian | 8 | 8 | 16
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 18 | 19 | 37
    White | 48 | 42 | 90
    More than one race | 5 | 5 | 10
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity. The number of participants represents those who provided data for this outcome measure.
  Participants
    Hispanic or Latino | 32 | 30 | 62
    Not Hispanic or Latino | 51 | 49 | 100
    Unknown or Not Reported | 0 | 0 | 0
Current Student [Count of Participants; unit: Participants] — Current Student. The number of participants represents those who provided data for this outcome measure.
  Participants | 45 | 41 | 86

OUTCOME MEASURES:

1. Primary Outcome: Typical Number of Drinks Per Occasion
Description: Measures the typical number of drinks consumed per occasion.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Typical number of drinks per occasion
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 77 | 75
Typical number of drinks per occasion | 3.75 (2.857) | 3.67 (3.027)

2. Primary Outcome: Typical Number of Drinks Per Occasion
Description: Measures the typical number of drinks consumed per occasion.
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Typical number of drinks per occasion
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 72 | 73
Typical number of drinks per occasion | 2.85 (2.396) | 3.05 (3.027)

3. Primary Outcome: Young Adult Alcohol Consequences Questionnaire
Description: The Young Adult Alcohol Consequences Questionnaire will asses consequences from drinking.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of Consequences
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 77 | 75
Number of Consequences | 9.66 (5.92) | 8.80 (6.37)

4. Primary Outcome: Young Adult Alcohol Consequences Questionnaire
Description: The Young Adult Alcohol Consequences Questionnaire will asses consequences from drinking.
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of Consequences
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 73 | 72
Number of Consequences | 5.97 (6.07) | 5.78 (6.37)

5. Primary Outcome: Alcohol Protective Behavioral Strategies
Description: Alcohol Protective Behavioral Strategies (i.e., tips and strategies used to reduce harm when drinking) will be assessed with the Protective Behavioral Strategies Survey-20. Protective Behavioral Strategies were assessed using the full Protective Behavioral Strategies Scale-20 (PBSS-20), which measures the frequency of using strategies to limit alcohol use and related consequences. The PBSS-20 consists of 20 items rated on a 6-point Likert-type scale (1 = Never to 6 = Always). Scores are averaged across items, with higher values indicating greater use of protective behavioral strategies (i.e., a more favorable outcome).
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a 1-6 scale
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 75 | 74
Units on a 1-6 scale | 3.67 (.706) | 3.63 (.867)

6. Primary Outcome: Alcohol Protective Behavioral Strategies
Description: as for outcome 5
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a 1-6 scale
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 72 | 71
Units on a 1-6 scale | 3.83 (.878) | 3.78 (1.059)

7. Primary Outcome: Average Days Cannabis Use Past Two Months
Description: This measure will assess typical days cannabis was used the past two months.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Average days cannabis use past two month
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 76 | 75
Average days cannabis use past two month | 5.74 (3.01) | 6.09 (3.15)

8. Primary Outcome: Average Days Cannabis Use Past Two Months
Description: This measure will assess typical days cannabis was used the past two months.
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Average days cannabis use past two month
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 72 | 73
Average days cannabis use past two month | 4.46 (3.42) | 4.60 (3.06)

9. Primary Outcome: Cannabis Protective Behavioral Strategies
Description: Cannabis Protective Behavioral Strategies were assessed using the Protective Behavioral Strategies for Marijuana Scale, a 26-item measure evaluating the frequency of strategies used to reduce cannabis use and related harm. Items are rated on a 6-point Likert scale (1 = Never to 6 = Always). Scores are averaged across items, with higher scores indicating greater use of protective behavioral strategies (i.e., a more favorable outcome).
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a 1-6 scale
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 75 | 74
Units on a 1-6 scale | 3.20 (.677) | 3.22 (.985)

10. Primary Outcome: Cannabis Protective Behavioral Strategies
Description: as for outcome 9
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a 1-6 scale
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 71 | 71
Units on a 1-6 scale | 3.56 (1.03) | 3.61 (1.23)

11. Primary Outcome: Marijuana Consequences Questionnaire
Description: The Marijuana Consequences Questionnaire and a modified version will measure a broad range of negative cannabis consequences.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of cannabis consequences
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 76 | 74
Number of cannabis consequences | 28.16 (16.41) | 28.83 (20.73)

12. Primary Outcome: Marijuana Consequences Questionnaire
Description: as for outcome 11
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of cannabis consequences
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 73 | 71
Number of cannabis consequences | 20.76 (20.34) | 21.38 (18.20)

13. Primary Outcome: Simultaneous Alcohol and Marijuana Use
Description: Questions regarding SAM use will be adapted from MTF.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of times SAM use past two months
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 75 | 75
Number of times SAM use past two months | .93 (.251) | .93 (.250)

14. Primary Outcome: Simultaneous Alcohol and Marijuana Use
Description: Questions regarding SAM use will be adapted from MTF.
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of times SAM use past two months
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 74 | 71
Number of times SAM use past two months | .88 (.332) | .83 (.377)

15. Primary Outcome: Feasibility- Number of Participants Who Visited the Online Intervention
Description: The Number of Participants who Visited the Online Intervention
Time Frame: 2 Month
Population: The number of participants represents those who provided data for this outcome measure. Only the intervention group was assessed.
Measure: Number; unit: Participants
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 78 | 0
Participants | 78 |

16. Primary Outcome: Feasibility- Number of Online Modules Selected
Description: The number of modules participants in the intervention condition selected to view.
Time Frame: Baseline
Population: The number of participants represents those who provided data for this outcome measure. Only the intervention group completed this measure.
Measure: Mean (Standard Deviation); unit: Mean modules selected
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 78 | 0
Mean modules selected | 8.80 (2.80) |

17. Primary Outcome: Acceptability- System Usability Scale
Description: Scores on a measure of subjective assessments of usability (SUS) from participants in the intervention condition. Total score from 0 to 100 with higher scores indicating higher usability.
Time Frame: Post-Intervention
Population: The number of participants represents those who provided data for this outcome measure. Only the intervention group completed this measure. The control group did not receive this measure.
Measure: Mean (Standard Deviation); unit: Mean SUS score
Arm/Group | Online and Text Message Intervention | Assessment Only Control
Number analyzed (Participants) | 78 | 0
Mean SUS score | 76.60 (13.20) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial screening and final follow-up for each participant, a period of approximately 2 months.
Description: We used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | Online and Text Message Intervention | Assessment Only Control
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/79
Other Adverse Events (participants affected / at risk) | 0/83 | 0/79

LIMITATIONS AND CAVEATS:
This is a small pilot trial designed to collect feasibility and acceptability information. All findings are based on self-report of alcohol and cannabis use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04978129/Prot_SAP_000.pdf